CLINICAL TRIAL: NCT05228067
Title: Enhancing Brain Health to Prevent Type 2 Diabetes
Brief Title: Enhancing Brain Health by TDCS in Persons with Overweight and Obesity
Acronym: STIM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 172/2021BO1
Record Dates: First submitted 2021-11-12; First posted 2022-02-08 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Insulin Resistance; Obesity; Diabetes Type 2
Keywords: tDCS; MRI; hypothalamus; functional connectivity
MeSH Terms: conditions — Insulin Resistance; Obesity; Diabetes Mellitus, Type 2 | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: All participants receive sham stimulation, anodal stimulation and cathodal stimulation in a pseudo-randomized order on three separate measurement days.
Who Masked: Participant, Investigator
Masking Description: Stimulation protocol is applied in a double blind fashion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Anodal stimulation (Active Comparator): Anodal tDCS of the hypothalamus network
  Interventions: Device: anodal transcranial direct current stimulation
- Cathodal stimulation (Active Comparator): Cathodal tDCS of the hypothalamus network
  Interventions: Device: cathodal transcranial direct current stimulation
- Sham stimulation (Sham Comparator): Sham tDCS of the hypothalamus network
  Interventions: Device: sham transcranial direct current stimulation

INTERVENTIONS:
Device: anodal transcranial direct current stimulation — anodal tDCS of the hypothalamus resting-state functional connectivity network using 12 Electrodes of the Starstim device by Neuroelectrics. The total injected current will never go beyond 4 milliamp, which will be split among the different stimulation electrodes.
  Other Names: anodal tDCS; excitatory tDCS
  Arms: Anodal stimulation
Device: cathodal transcranial direct current stimulation — anodal tDCS of the hypothalamus resting-state functional connectivity network using 12 Electrodes of the Starstim device by Neuroelectrics. The total injected current will never go beyond 4 milliamp, which will be split among the different stimulation electrodes.
  Other Names: cathodal tDCS; inhibitory tDCS
  Arms: Cathodal stimulation
Device: sham transcranial direct current stimulation — Double blind sham stimulation of the hypothalamus resting-state functional connectivity network (ramp-up ramp-down stimulation will be applied for 30 seconds)
  Other Names: sham tDCS
  Arms: Sham stimulation

SUMMARY:
Disturbances in the hypothalamus communication pathways with other regions in the brain and the periphery may represent a potential link between metabolic and cognitive health. The current project evaluates whether enhancing synaptic plasticity of this pathway can improve weight management, insulin sensitivity, and cognitive functions. In recent studies, we were able to show that the human brain is sensitive to insulin with favorable effects on peripheral metabolism and cognition. These brain regions encompass the hypothalamus and its connections to the striatum and prefrontal cortex. We want to investigate whether it is possible to enhance neuroplasticity of insulin-responsive brain regions to suppress the weight gain trajectory and improve dopamine-dependent cognitive functions in people with a high risk to develop type 2 diabetes. For this purpose, neuroimaging tools using high-definition transcranial direct current stimulation (HD-tDCS) and magnetic resonance imaging (MRI) will be implemented to assess synaptic plasticity of a neural network essential for metabolic and cognitive health.

DETAILED DESCRIPTION:
The overarching aim of the study is to investigate the possibility to enhance neuroplasticity of the hypothalamus network to improve metabolism and dopamine-dependent cognitive functions.

Specific objectives

* Specifically, it is the first aim to study the predictive value of white matter microstructure (fiber tracts structurally connecting the target network) for tDCS-intervention response and to investigate tDCS-induced neuroplasticity changes of the hypothalamus brain network using functional magnetic resonance imaging (fMRI).
* It is the second aim of this study to deepen our understanding of brain structure and function of the target network, which is known to rely on the neurotransmitter dopamine for its communication. Hence, we will use dopamine-dependent cognitive and eating behavior assessments.

Participants will receive a thorough screening to obtain body composition by MRI, anthropometric measures, fasting glucose and insulin, indirect calorimetry, and general cognitive functions. Thereafter, participants will participate in three measurement days (separated by approx. one week) to receive a 25 min tDCS stimulation targeting the hypothalamus network in a double-blind cluster-randomized. Participant are randomized on three conditions: sham stimulation, anodal and cathodal stimulation. During the non-invasive brain stimulation, participants will perform a stop-signal task. On each measurement day, structural and functional MRI measurements are performed before and after stimulation. Dopamine-dependent behavior (i.e. reward task) will be assessed during fMRI measurement. Subsequently, participants will receive a breakfast buffet. The caloric intake from fat, carbohydrates and protein will be documented. Subjective feeling of hunger and food craving will be assessed using a visual analogue scale before stimulation, directly after stimulation and after breakfast. Food pictures will be rated on a laptop for taste and healthiness.

ELIGIBILITY:
Inclusion Criteria:

* Written consent to participate in the study
* Written consent to be informed about incidental findings

Overweight and obese participants:

* Body mass index (BMI) between 28 and 39.5 kg/m2
* Age between 20 to 65 years of age
* Waist circumference > 80 cm for women, > 94 cm for men

Sex and age matched normal weight individuals:

* Body mass index (BMI) between 19.5 and 24.5 kg/m2
* Age between 20 to 65 years of age

Exclusion Criteria:

* Insufficient knowledge of the German language
* Persons who cannot legally give consent
* Pregnancy or lactation
* History of severe mental or somatic disorders including neurological diseases (incl. Epileptic seizures)
* Taking psychotropic drugs
* Previous bariatric surgery
* Acute infection within the last 4 weeks
* Hemoglobin values less than 12g/dl for women, less than 14 g/dl for men
* Current participation in a lifestyle intervention study or a pharmaceutical study
* Contradictions to a MRI measurement (e.g. metal implants)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-08 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in neuroplasticity | 20 minutes directly before and after tDCS stimulation
  Fractional anisotropy (FA) of the target network
Change in functional connectivity | 20 minutes directly before and after tDCS stimulation
  Resting state functional connectivity of the target network
Change in eating behavior | 1 hour after tDCS stimulation
  Caloric intake (kcal), Free-choice, ad libitum food intake from a standardized breakfast buffet. The caloric intake from fat, carbohydrates and protein will be documented
Change in dopamine-dependent cognitive function | 20 minutes after tDCS stimulation
  Changes in dopamine-dependent cognitive function and reward sensitivity measured by a reward-based decision-making task

SECONDARY OUTCOMES:
Change in subjective ratings | 5 minutes before tDCS stimulation, 5 minutes after tDCS stimulation and 5 minutes after buffet
  Change in subjective ratings will be assessed using a visual analogue scale for hunger and subjective feeling of craving using a questionnaire (Food craving questionnaire). Visual analogue scale using a range from 0 to 10 cm, higher values indicating more hunger. Food craving questionnaire based on ordinal scale from 1 to 5, higher values indicating more food craving
Performance during stop-signal task | task is performed during 25-minutes tDCS stimulation
  Outcome measures cover direction errors, proportion of successful stops, reaction time on Go trials, and stop signal reaction time (SSRT)
Tastiness and healthiness rating of food stimuli | task is performed immediately after buffet
  Using a computer based task, participants rate food pictures of low caloric and high caloric foods and snacks on a 5-point scale based on subjective tastiness and healthiness
Food choice | task is performed immediately after buffet
  Using a computer based task, participants have to choose food items they preferred to eat compared to a reference food on a 5-point choice scale. The reference (or "neutral") food item is individually determined based the health and taste rating [Scale: 1= not tasty/ not healthy up to 5= very tasty/ very healthy]

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No